CLINICAL TRIAL: NCT02184884
Title: Effect of Perioperative Clopidogrel Responsiveness on Ischemic Outcome in Patients With Acute Coronary Syndrome Undergoing Off-pump Coronary Artery Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0172
Record Dates: First submitted 2014-06-30; First posted 2014-07-09 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: off-pump coronary artery bypass surgery, clopidogrel responsiveness, ischemic outcome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MACE group: the patients with MACE after OPCAB
  Interventions: Device: MACE after OPCAB
- no MACE group: the patients without MACE after OPCAB
  Interventions: Device: without MACE after OPCAB

INTERVENTIONS:
Device: MACE after OPCAB
  Groups: MACE group
Device: without MACE after OPCAB
  Groups: no MACE group

SUMMARY:
The whole blood Thrombelastograph (TEG®) Platelet Mapping™ assay measures clot strength, maximal amplitude (MA), reflecting maximal platelet function, and detects the reduction in platelet function, presented as percentage inhibition, by both aspirin and clopidogrel. A study reported that the TEG® can be used as routine monitoring of the variability in ADP receptor inhibition and of antiplatelet therapy. Therefore, using TEG Platelet Mapping assay, we could find out the perioperative clopidogrel responsiveness of the patients with ACS undergoing OPCAB.

The purpose of this study is to determine whether the rate of the major adverse cardiac events (MACE, a combined endpoint of MI, revascularization and cardiac death) is higher in the patients with high degree of clopidogrel resistance, who are scheduled to undergo the OPCAB due to ACS.

ELIGIBILITY:
Inclusion Criteria:

1. the patients with ACS undergoing OPCAB
2. the patients over 20 years of age
3. the patient who have been taking [100 mg of Aspirin] and [75 mg of clopidogrel or 180 mg of ticagrelor] for more than one week and who continue within 3 to 5 days prior to surgery

Exclusion Criteria:

1. re-operation or emergency operation
2. the patients with bleeding tendency of decreased liver function
3. Left ventricular ejection fraction < 40% by echo
4. preoperative hematocrit < 33% or platelet count < 100,000/mm3 or creatinine > 1.4 mg/dL
5. abnormal preoperative prothrombin time or activated partial thromboplastin time
6. preoperative use of other PO antiplatelet drugs or PO anticoagulants

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute coronary syndrome (ACS) undergoing off-pump coronary artery bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Rate of the major adverse cardiac events | at 30 days after surgery
  major adverse cardiac events(MACE) includes the MI, revascularization and cardiac death. Rate of the MACE will be higher in the patients with high degree of clopidogrel resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Soh S, Shin YR, Song JW, Choi JH, Kwak YL, Shim JK. Platelet Reactivity and Outcomes after Off-Pump Coronary Surgery in Acute Coronary Syndrome Patients. J Clin Med. 2022 Jun 8;11(12):3285. doi: 10.3390/jcm11123285. PMID 35743360